CLINICAL TRIAL: NCT04001959
Title: Comparison of the Potential for Dentine Discoloration of Silver Diamino Fluoride and Silver Diamino Fluoride Associated With Potassium Iodide
Brief Title: Potential for Dentine Discoloration of Silver Diamino Fluoride Associated With Potassium Iodide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of the Valleys of Jequitinhonha and Mucuri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04243718.0.0000.5108
Record Dates: First submitted 2019-06-24; First posted 2019-06-28 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Dental Caries in Children
Keywords: Carostats; Clinical trial; Preventive dentistry; Preschoolers
MeSH Terms: interventions — silver diamine fluoride; Potassium Iodide

STUDY DESIGN:
Intervention Model Description: A randomized, controlled study in which the variables were evaluated 1 week, 15 days, 1 and 2 months after the intervention. For the allocation of participants, a Randomization ratio of 1: 1 was performed.
Who Masked: Participant, Care Provider
Masking Description: Single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silver Diamine Fluoride (Active Comparator): Initially a prophylaxis will be done on the tooth to be treated with Robinson brush and prophylactic paste and then the relative isolation (with mouth openers and cotton rollers) and protection of the soft tissues with vaseline in the region to be treated to protect the surrounding tissues will be carried out. Next, dry the tooth for 30 seconds with air jet followed by a drop of 30% Diamino Fluoride Silver with a disposable applicator brush for 3 minutes and after that time washing for 1 minute.
  Interventions: Procedure: Silver Diamine Fluoride with Potassium Iodide
- Silver Diamine Fluoride with Potassium Iodide (Experimental): Initially a prophylaxis will be done on the tooth to be treated with Robinson brush and prophylactic paste and then the relative isolation (with mouth openers and cotton rollers) and protection of the soft tissues with vaseline in the region to be treated to protect the surrounding tissues will be carried out. Then the tooth is dried for 30 seconds with an air jet and applied one drop of the Diamino 30% Silver Fluoride with a disposable applicator brush for 3 minutes and one drop of potassium iodide solution immediately on the surface treated with Diamino , until the formed creamy white color becomes transparent. After these steps have been completed, rinse with water for 1 minute.
  Interventions: Procedure: Silver Diamine Fluoride with Potassium Iodide

INTERVENTIONS:
Procedure: Silver Diamine Fluoride with Potassium Iodide — Dry the tooth for 30 seconds with air jet and apply one drop of Diamino 30% Silver Fluoride with a disposable applicator brush for 3 minutes and one drop of potassium iodide solution immediately on the treated surface, then wash.

SUMMARY:
The objective of this randomized clinical trial will be the comparison of dentine discoloration after treatment with: Silver Diamino Fluoride and Silver Diamino Fluoride associated with Potassium Iodide for caries lesions in posterior primary teeth. The study sample will consist of children presenting caries lesion in dentin, without reporting spontaneous pain. The children will be allocated into 2 groups that will correspond to the treatments with the use of SDF (Group 1), SDF + PI (Group 2). Treatment will be performed by trained and calibrated researchers. Examiners will be blind to the treatment received. Initially, data will be collected on socio-demographic aspects, characteristics of children, and clinical aspects. Clinical, photographic and initial evaluations will be performed after 1 week, 15 days, 1 and 2 months after treatment. The results obtained will be typed and organized in a database, using the software Statistical Package for Social Science (SPSS), version 22.0 and descriptive, bivariate analyzes will be performed.

DETAILED DESCRIPTION:
Primary Objective:

To compare dentine discoloration in caries lesions in the deciduous dentition after Silver Diamino Fluoride treatment with and without association with Potassium Iodide (PI).

Secondary Objective:

To compare the effectiveness of the methods in the inactivation of active carious lesions Compare the inactivation time of the lesions between the groups Compare the presence of biofilm accumulation in the different comparing the differences in the effectiveness of the methods for inactivation of lesions on different surfaces.

Scratchs:

The risks inherent to the study are related to the embarrassment at the moment of answering the questionnaires, however they will be carried out in a reserved space. There is a risk of discomfort for the child or the caretaker during the evaluation and / or clinical examination. However, the examiners will be prepared to identify any possible discomfort and discontinue the evaluation if this occurs. The risks may also be related to the identification of the participants, however the medical record with questionnaires will only be accessed by the research team. There are also clinical risks inherent in the progression of caries, in which case the team will perform conventional and indicated the current clinical situation (restoration, endodontics, dental extraction). The research will be immediately suspended if there is suspicion of any risk or damage to the health of the participant.

Benefits:

The benefits relate to remission of signs and symptoms after treatment. In addition, there will be maintenance of the dental elements in the oral cavity of the child until its physiological exfoliation, thus avoiding the damages resulting from the early loss of a deciduous tooth such as: reduction in mastication and phonetic efficiency, loss of vertical dimension, impairment of aesthetics , installation of deleterious oral habits, impairment of craniofacial development, damage to the permanent dentition, and intense psychological repercussions.

Proposed Methodology:

Ten children will be examined by the examiner and an experienced investigator in order to obtain inter-examiner agreement. The sequence of procedures to be performed in the participants during the study will be: 1st Consultation: Application of the sociodemographic, general health of the child and habits questionnaire; biofilm evaluation; Clinical evaluation of the caries (ICDAS + AAL); Photograph of the lesion; Behavioral evaluation of the child; Application of treatment (Randomization). 2nd Consultation (1 week): Photography; Pain evaluation (DDQ-B), behavioral evaluation. 3rd Consultation (15 days): Photography; Treatment follow-up; Pain evaluation (DDQ-B); Behavioral evaluation of the child.4ª Consultation (1 month): Photography; Biofilm evaluation; Treatment follow-up; Pain evaluation (DDQ-B); Behavioral evaluation of the child. 5th Consultation (2 months): Photography; Biofilm evaluation; treatment follow-up; Pain evaluation (DDQ-B); Clinical evaluation of caries lesion (ICDAS + AAL); Behavioral assessment of the child. Children of the study, their parents and the examiner will remain blind to the allocation of the children's group. Blinding of the operator will not be possible, since the technique of use allows the identification of the material used.

Data Analysis Methodology:

The results obtained will be typed and organized in a database, using the software Statistical Package for Social Science (SPSS), version 22.0. Initially, a description of the absolute and relative frequencies will be performed, as well as the measures of central tendency of the variables studied. In addition, the distribution of the data will be verified in order to evaluate if the data present normality, which will guide the choice by the use of parametric or non-parametric tests. Bivariate analysis will be performed to verify the association between the dependent variables and the type of treatment. The categorical variables will be evaluated using Fisher's Qui-square and Exact tests. For the quantitative variables, the study of the distribution of the data will initially be performed. If these present a normal distribution, the Anova parametric tests and paired T-test will be used. If the distribution is not normal, the Friedman and Wilcoxon tests will be used. The null hypothesis is that there is no association between the variables (p> 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Children who have at least one vital deciduous tooth with a dentin cavitated lesion.
* Children whose parents / guardians agree to their child's participation in the study.

Exclusion Criteria:

* Child with systemic health impairment;
* Child who has already performed dental treatment on the tooth to be included in the research;
* Sensitivity to chemicals used;
* Tooth with spontaneous pain;
* Tooth with pulp wrapping;
* Radiographic evidence of pathological internal or external resorption of the root;
* Radiographic evidence of periapical lesion;

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Dentin color change | 1 week, 15 days, 1 and 2 months
  In all the consultations will be made photographic shoots of the tooth with purpose of comparison. Then all images will be downloaded to the computer and analyzed using the Windows program - Paint. The tooth will be analyzed on all its faces. The coloration will be evaluated in scores from 0 to 4 where 0 is white, 1 yellow, 2 light brown, 3 dark brown and 4 black.

SECONDARY OUTCOMES:
Clinical success based on the International System for Assessment and Detection of Caries (ICDAS) | 1 and 2 months
  The ICDAS describes six stages of dental caries extension, ranging from initial visible changes in the enamel to the sharp dentin cavitation. We will use this index to evaluate the stoppage and prevention of caries by the proposed treatment.
Parental Satisfaction Scale | 1 and 2 months
  Satisfaction with the type of treatment proposed. Scale ranging from 0 to 10, where 0 is the worst condition and 10 is the best condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Priscila Seixas Mourão, Diamantina, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No